CLINICAL TRIAL: NCT01701479
Title: A Phase I/II Dose Schedule Finding Study of ch14.18/CHO Continuous Infusion Combined With Subcutaneous Aldesleukin (IL-2) in Patients With Primary Refractory or Relapsed Neuroblastoma
Brief Title: Long Term Continuous Infusion ch14.18/CHO Plus s.c. Aldesleukin (IL-2)
Acronym: LTI
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: St. Anna Kinderkrebsforschung (Other)
Collaborators: University Medicine Greifswald (Other); St. Anna Children's Hospital, Vienna (Unknown); Hospital Universitario La Fe (Other); Istituto Giannina Gaslini (Other); Gustave Roussy, Cancer Campus, Grand Paris (Other); Schneider Children's Medical Center, Israel (Other); Great Ormond Street Hospital for Children NHS Foundation Trust (Other); University Hospital, Toulouse (Other); Johann Wolfgang Goethe University Hospital (Other); Jena University Hospital (Other); Children's University Hospital, Ireland (Other); University Hospital Tuebingen (Other); Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other); Alder Hey Children's NHS Foundation Trust (Other); University Hospitals Bristol and Weston NHS Foundation Trust (Other); Newcastle-upon-Tyne Hospitals NHS Trust (Other); The Leeds Teaching Hospitals NHS Trust (Other); NHS Greater Glasgow and Clyde (Other); Medical University of Graz (Other); Medical University Innsbruck (Other); Centre Leon Berard (Other); Hospital Infantil Universitario Niño Jesús, Madrid, Spain (Other); University Hospital Southampton NHS Foundation Trust (Other); Institut Curie (Other); Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 012010; 2009-018077-31 (EudraCT Number)
Record Dates: First submitted 2012-10-03; First posted 2012-10-05 (Estimated); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Neuroblastoma
Keywords: Neuroblastoma; Refractory neuroblastoma; Relapsed neuroblastoma; ch14.18/CHO; Aldesleukin (IL-2)
MeSH Terms: conditions — Neuroblastoma | interventions — aldesleukin; Interleukin-2; Isotretinoin

STUDY DESIGN:
Intervention Model Description: The patients will be randomised to immunotherapy with isotretinoin (13-cis-RA) and ch14.18/CHO, with or without aldesleukin (IL-2).
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental arm (Experimental): Subcutaneous aldesleukin (IL-2) will be given at a dose of 6 x 106 IU/m2/day in two 5 day blocks (days 1-5 and 8-12).
  A continuous infusion of ch14.18/CHO is started on day 8. The duration of the infusion is dependent on the assigned infusion schedule. The duration will range from 10 to 21 days. Three dose levels will be considered with respect to daily dose (7 mg/m2, 10 mg/m2, 15 mg/m2), which relates to total doses of 100 mg/m2,150 mg/m2 and 210 mg/m2.
  Patients will receive isotretinoin (13-cis-RA) 160 mg/m²/day divided into two equal doses given orally twice a day for 14 days after the completion of the ch14.18/CHO infusion. The starting day is dependent on the duration of ch14.18/CHO infusion and may be either day 19, 23, 24 or 30.
  Interventions: Drug: ch14.18/CHO; Drug: Aldesleukin; Drug: Isotretinoin
- Comparator arm (Active Comparator): A continuous infusion of ch14.18/CHO is started on day 8. The duration of the infusion is dependent on the assigned infusion schedule. The duration will range from 10 to 21 days. Three dose levels will be considered with respect to daily dose (7 mg/m2, 10 mg/m2, 15 mg/m2), which relates to total doses of 100 mg/m2,150 mg/m2 and 210 mg/m2.
  Patients will receive isotretinoin (13-cis-RA) 160 mg/m²/day divided into two equal doses given orally twice a day for 14 days after the completion of the ch14.18/CHO infusion. The starting day is dependent on the duration of ch14.18/CHO infusion and may be either day 19, 23, 24 or 30.
  Interventions: Drug: ch14.18/CHO; Drug: Isotretinoin

INTERVENTIONS:
Drug: ch14.18/CHO
  Other Names: Chimeric 14.18 anti-GD2 monoclonal antibody produced in Chinese hamster ovary cells
Drug: Aldesleukin
  Other Names: Proleukin; Interleukin-2; IL-2
  Arms: Experimental arm
Drug: Isotretinoin
  Other Names: 13-cis-Retinoic acid; 13-cis-RA

SUMMARY:
The main aim of this clinical trial is to find a way of giving ch14.18/CHO, in combination with subcutaneous aldesleukin (IL-2) and oral isotretinoin (13-cis-RA), to children and young people with primary refractory or relapsed neuroblastoma without intravenous morphine.

DETAILED DESCRIPTION:
Although a lot of children and young people with neuroblastoma can be cured with current standard chemotherapy, sometimes, particularly at relapse the disease no longer responds to standard drugs. Therefore, there is a need to find new drug combinations which will act against neuroblastoma which no longer responds to standard drugs.

Ch14.18/CHO has been shown to improve the outcome of patients with neuroblastoma. However, one of the side effects of receiving ch14.18/CHO is severe pain. High doses of intravenous morphine are needed to control the pain and this means that patients must stay in hospital. Results from other clinical trials have shown that giving ch14.18/CHO over a longer time reduces pain, yet the drug still works just as well to fight the neuroblastoma. The clinical trial aims to give ch14.18/CHO over a longer time so that intravenous morphine is not needed and that this treatment regimen can ultimately be given in an outpatient setting.

Ch14.18/CHO is a monoclonal antibody. Monoclonal antibodies are made in the laboratory and are designed to bind to specific cancer cells. Ch14.18/CHO was designed to bind to neuroblastoma cells and other cancer cells that express the GD-2 antigen. The GD-2 antigen is expressed by virtually all neuroblastoma cells. An antigen is a substance that stimulates an immune response in the body by producing antibodies. Thus, when ch14.18/CHO binds to the neuroblastoma cells, the body's immune system is stimulated to attack and kill the neuroblastoma cells. Ch14.18/CHO is called chimeric, because it was genetically engineered to consist of 30% mouse-protein and of 70% human protein.

Ch14.18/CHO represents a new kind of cancer therapy that, unlike chemotherapy and radiation, targets the destruction of cancer cells without destroying nearby healthy cells. There is laboratory evidence to suggest that ch14.18/CHO can activate the body's own immune cells to destroy cancer cells. These immune cells include killer cells that are activated or stimulated by aldesleukin (IL-2). Therefore this treatment is a combination of ch14.18/CHO and aldesleukin (IL-2).

Aldesleukin (IL-2) is a substance that is similar to a substance made by the body in all individuals. Under normal circumstances, the body makes small amounts of aldesleukin (IL-2) that help white blood cells fight infection. It is now possible to make aldesleukin (IL-2) in the laboratory and give humans much higher doses than their own body makes. There is evidence in the laboratory and in animals that aldesleukin (IL-2) increases the anti-cancer effect of monoclonal antibodies like ch14.18/CHO. We wish to study whether aldesleukin (IL-2) can help improve the effectiveness of ch14.18/CHO in humans.

In addition to ch14.18/CHO and aldesleukin (IL-2), isotretinoin (13-cis-RA) will also be given. Isotretinoin (13-cis-RA) is considered standard treatment for patients with neuroblastoma and works by induction of neuroblastoma cell death.

ELIGIBILITY:
Inclusion Criteria:

* At study entry patients must be > 1 year but <= 21 years of age. NOTE: Patients >21 years but <= 45 years of age, fulfilling the remaining criteria, may be enrolled in the study. These patients will be analysed separately and will not be included in the dose finding schedule algorithm. The purpose for inclusion of the older patients is to enable the collection of tolerability data.
* Patients must be diagnosed with neuroblastoma according to the INSS criteria.
* Must have received at least one previous high dose treatment followed by stem cell rescue after conventional therapy.
* Must fulfil one of the following criteria:
* Patients with stage 4 neuroblastoma on the current high-risk SIOPEN trial (HR-NBL-1/SIOPEN) either with primary refractory disease having had more than two front-line treatments or patients ineligible for the R2 randomization due to major delays after completed high-dose treatments.
* Treated and responding relapse after primary stage 4 disease, without signs of progression at study entry
* Treated and responding disseminated relapse after primary localized neuroblastoma without signs of progression at study entry.
* Patients must have a performance status greater or equal 70% (Lansky Score or Karnofsky, see Appendix 1: performance Scales , page 91)
* Patients must have an estimated life expectancy of at least 12 weeks.
* Patients must consent to the placement of a central venous line, if one has not already been placed.
* Patients must be off any standard or experimental treatments for at least two weeks prior to study entry and be fully recovered from the short term major toxic effects.
* Patients must have no immediate requirements for palliative chemotherapy, radiotherapy or surgery.
* At least 4 weeks after major surgery (e.g. laporotomy or thoracotomy) and fully recovered from any post-surgical complications.
* HIV and Hepatitis B negative.
* Females of childbearing potential must have a negative pregnancy test. Patients of childbearing potential must agree to use an effective birth control method. Female patients who are lactating must agree to stop breast-feeding.
* Patients may have had prior CNS metastasis providing the following criteria are all met:
* the patient's CNS disease has been previously treated,
* the patient's CNS disease has been clinically stable for four weeks prior to starting this study (assessment must be made clinically and by CT or MRI scan),
* the patient is off steroids for CNS disease for four weeks prior to starting on study and during the course of the study.
* Patients with seizure disorders may be enrolled if on anticonvulsants and are well controlled.
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional and national requirements for human studies must be met.
* Laboratory Testing:
* Patients should have a shortening fraction of >= 30 % by Echocardiogram.
* Patients should have FEV1 and FVC >60% of the predicted by pulmonary function tests. Children unable to do PFTs should have no dyspnea at rest and a pulse oximetry >94% on room air.
* All patients must have adequate bone marrow function as defined by ANC >1 10^9/L, platelets >= 50 10^9/L and haemoglobin > 9.0 g/dL.
* Patients must have adequate liver function, as defined by an ALT or AST < 5 x normal and a total bilirubin < 1.0 mg/dL.
* Patients must have adequate renal function, as defined by a serum creatinine <1.5 mg/dL or a creatinine clearance or radioisotope GFR of > 60 mL/minute/1.73m2.

Exclusion Criteria:

* Patients with progressive disease
* Patients who have previously received treatment with ch14.18/SP2/0 and/or ch14.18/CHO.
* Platelet transfusion dependent.
* Patients with significant intercurrent illnesses and/or any of the following:
* Patients with symptoms of congestive heart failure or uncontrolled cardiac rhythm disturbance.
* Patients with significant psychiatric disabilities or uncontrolled seizure disorders.
* Patients with active infections.
* Patients with a clinically significant neurologic deficit or objective peripheral neuropathy (Grade >2) are ineligible.
* Patients with clinically significant, symptomatic, pleural effusions.
* Patients who require, or are likely to require, corticosteroid or other immunosuppressive drugs.
* Concurrent treatment with any non-trial anticancer therapies.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 288 (Estimated)
Dates: Start 2012-01; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Event free survival | through study completion, an average of 1 year
  The primary endpoint is event free survival calculated from the date of randomisation. The following will be considered as events:
  * disease progression or relapse
  * death from any cause
  * second neoplasm

SECONDARY OUTCOMES:
Pain-toxicity endpoint | through study completion, an average of 1 year
  assessment of pain intensity and relief by appropriate medication with a validated self-report tool (Wong-Baker Faces Pain Rating Scale, FPS-R)
Efficacy endpoint | through study completion, an average of 1 year
  validation of the correlation between activated NK cells and ch14.18/CHO level with ADCC by using serum and MNC from patients
Systemic immune modulation/response | through study completion, an average of 1 year
  repeated analysis of NK-cell activation, soluble IL-2 receptor, ADCC, CDC and anti-idiotype response (HAMA and HACA)
Assessment of absolute lymphocyte counts and absolute NK cell numbers after the respective cycles as a measurement of response to s.c. aldesleukin (IL-2) in the standard treatment arm. | through study completion, an average of 1 year
Determination of pharmacokinetics of ch14.18/CHO by assessing blood levels of ch14.18/CHO via ELISA (Enzyme-linked-Immunosorbent Assay) | through study completion, an average of 1 year
  determination of the pharmacokinetics of ch14.18/CHO (ELISA analysis of ch14.18/CHO blood levels)
Evaluation of anti-tumour response in patients with measureable disease | through study completion, an average of 1 year
  Bone marrow, skeletal lesions, soft tissue lesions, lymph nodes and/or primary tumour site as measured by immunocytology, mIBG, CT and/or MRI
Evaluation of impact of KIR/KIRL mismatch and Fc receptor polymorphisms on EFS (PCR sequence-specific primer technique) | through study completion, an average of 1 year
  Immunomodulation induced by the treatment will be complemented by a whole blood assay. Fc Receptor polymorphisms and KIR/KIR Ligand mismatch analysis will be done via KIR genotyping on patient DNA samples by PCR sequence-specific primer technique

CONTACTS AND LOCATIONS:
Overall Officials: Holger Lode, MD, PhD, Principal Investigator — University Medicine Greifswald
Locations (14):
- St. Anna Kinderspital, Vienna, Austria
- France (2):
  - Institut Curie, Paris
  - Institut Gustave Roussy, Villejuif
- University Children's Hospital, Greifswald, Germany
- Schneider Children's Medical Centre of Israel, Petach Tikvah, Israel
- Gaslini Children's Hospital, Genova, Italy
- Hospital Universitario La Fe, Valencia, Spain
- United Kingdom (7):
  - Birmingham Children's Hospital NHS Foundation Trust, Birmingham
  - University Hospitals Bristol NHS Foundation Trust, Bristol
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - Alder Hey Children's NHS Foundation Trust, Liverpool
  - University College Hospitals NHS Foundation Trust, London
  - Great Ormond Street Hospital for Children NHS Foundation Trust, London
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle

REFERENCES:
- See also: Related Info — http://www.kinderkrebsforschung.at/
- See also: Related Info — https://www.siopen-r-net.org/